CLINICAL TRIAL: NCT04046744
Title: Axillary Block in Association With Analgesic Truncal Blocks of the Median and Radial Nerves at the Elbow for Wrist Surgery.
Brief Title: Axillary Block in Association With Analgesic Truncal Blocks at the Elbow for Wrist Surgery.
Acronym: BAXASSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/03
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Wrist Fracture
Keywords: Regional anesthesia; Analgesia; Ultrasound
MeSH Terms: conditions — Wrist Fractures; Agnosia | interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAX (Active Comparator)
  Interventions: Procedure: Axillary brachial plexus block with a long-acting local anesthetic; Drug: Ropivacaine
- BAX-Asso (Experimental)
  Interventions: Procedure: Axillary brachial plexus block with a short-acting local anesthetic + Analgesic block at the elbow with a long-acting local anesthetic; Drug: Ropivacaine; Drug: Lidocaine

INTERVENTIONS:
Procedure: Axillary brachial plexus block with a long-acting local anesthetic — axillary block with 15-30 ml Ropivacaine 0,5%.
  Arms: BAX
Procedure: Axillary brachial plexus block with a short-acting local anesthetic + Analgesic block at the elbow with a long-acting local anesthetic — axillary block with 15-30 ml Lidocaine 1,5% + radial and medial nerve block at the elbow with 3-7 ml Ropivacaine 0,5%.
  Arms: BAX-Asso
Drug: Ropivacaine — axillary block with 15-30 ml Ropivacaine 0,5%
  Arms: BAX
Drug: Ropivacaine — radial and medial nerve block at the elbow with 3-7 ml Ropivacaine 0,5%
  Arms: BAX-Asso
Drug: Lidocaine — axillary block with 15-30 ml Lidocaine 1,5%
  Arms: BAX-Asso

SUMMARY:
Fractures of the forearm bones that occur around the wrist are common in the elderly. Standard anesthesia for its surgical treatment is regional anesthesia (RA): supraclavicular block, infraclavicular block or axillary block (BAX). However, these techniques have some limitations, such as the postoperative pain management and the non-specificity of the analgesia. Indeed analgesia is not specific to the wrist and extends to the elbow and forearm, preventing rapid recovery of elbow flexion and extension when a long-acting local anesthetic (LA) is used. Recently RA techniques associating proximal anesthetic blocks with distal analgesic blocks have been proposed to serve a dual objective: good anesthesia for surgery and specific analgesia.

The hypothesis of this study is that, for the wrist surgery, axillary block using a short-acting LA combined with analgesic blocks at the elbow using a long-acting LA could provide a RA installation time reduction, an optimal surgical comfort, a longer post-operative analgesia duration and a faster recovery from motor block.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, open-Label study compares two techniques :

* BAX (usual technique) : Axillary brachial plexus block (Axillary block) with a long-acting LA (Ropivacaine)
* BAX-Asso (experimental technique) : Axillary brachial plexus block (Axillary block) with a short-acting local anesthetic (Lidocaine) + Analgesic block at the elbow with a long-acting local anesthetic (Ropivacaine) Every block will be performed under Ultrasound. BAX will be performed using a multi-injection technique at contact with median (nM), radial (nR), ulnar (nU), musculocutaneous (nMC) and medial antebrachial cutaneous (nCMAB) nerves. 15-30 mL of LA will be injected.

Analgesic truncal blocks of the median and radial nerves will be performed at the elbow. 3-7 mL of LA will be injected.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing wrist fracture surgery under regional anesthesia
* Consent for participation
* Affiliation to the French social security system

Exclusion Criteria:

* Chronic use of opiod analgesics
* Chronic pain syndrome or fibromyalgia
* Contraindication for locoregional anesthesia
* Contraindication for opioid
* ASA IV
* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Level of pain when the patient recovers the flexion of the forearm on the arm | 24 hours
  Pain VRS ranging from 0 to 10 (0=no pain, 10=worst possible pain)

SECONDARY OUTCOMES:
Duration of motor block at the elbow | 24 hours
  Time between the performance of regional anesthesia and the elbow flexion recovery
Axillary block success | 40 minutes
  Assess of motor block and sensory perception to pin-prick in the distribution of the five terminal branches at 10, 20, and 30 minutes postinjection.
  Motor block: complete (2=paralysis), partial (1=paresis), or none (0). Motor function assessed in the following manner: wrist and finger flexion (median nerve), wrist and finger extension (radial nerve), thumb adduction and flexor carpi ulnaris flexion (ulnar nerve), and biceps flexion (musculocutaneous nerve).
  Sensory block: complete/anesthesia (2=loss of sensation to pinprick), partial/analgesia (1=dull sensation to pinprick), or none (0=sharp sensation to pinprick).
  Sensory distribution assessed in the following areas: thenar eminence and thumb tip (median nerve), dorsum of hand (radial nerve), fifth digit fingertip (ulnar nerve), lateral aspect of forearm (musculocutaneous nerve) and medial aspect of forearm (medial antebrachial cutaneous nerve).
  Successful blockade is defined by a sensory-motor score ≥ 3.
Feasibility of the wrist surgery | 2 hours
  Usage (or not) of an additional anesthetic procedure to perform the surgery
Duration of postoperative analgesia | 72 hours
  Time between the performance of regional anesthesia and the first dose of rescue analgesia with opioides.
Postoperative morphine consumption | 48 hours
  Cumulated dose of oxynorm (mg)
Sleep quality | Day 2 After Surgery
  Incidence of sleep disorders
Complications during block performance | 15 minutes
  Incidence of vascular puncture, paresthesia, intraneural injection and intravascular passage
Complications immediately after block | 2 hours
  Onset of vertigo, nausea or vomiting
Postoperative complications | Day 15 After Surgery
  Questionnaire about potential sensory anomalies such as numbness, itching or tingling

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Clinique du Pré, Le Mans, Pays de la Loire Region
  - Hôpital Privé Paul D'Egine, Champigny-sur-Marne, Île-de-France Region
  - CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region
  - Hôpital Privé Armand Brillard, Nogent-sur-Marne, Île-de-France Region
  - Clinique Bizet, Paris, Île-de-France Region
  - Clinique Jouvenet, Paris, Île-de-France Region
  - Clinique Rémusat, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No